CLINICAL TRIAL: NCT00437879
Title: Pilot Investigation of Ultrasound Imaging and Spectroscopy and Ultrasound Imaging of Vascular Blood Flow as Early Indicators of Breast Cancer Response to Neoadjuvant Treatment
Brief Title: Ultrasound Imaging, Spectroscopy and Ultrasound Imaging of Vascular Blood Flow as Early Indicators of Breast Cancer Response to Neoadjuvant Treatment.
Status: Recruiting | Type: Observational
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Gregory Czarnota, Dr., Sunnybrook Health Sciences Centre
Other Study IDs: 185-2006
Record Dates: First submitted 2007-02-20; First posted 2007-02-21 (Estimated); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Breast Cancer Invasive
Keywords: Breast Cancer; Ultrasound; Neoadjuvant Treatment
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
We have previously demonstrated that high-frequency ultrasound and spectroscopy, and recently conventional-frequency ultrasound and spectroscopy may be used to detect cell death in vitro, in situ and in vivo. The method can detect different forms of cell death and has been demonstrated to be sensitive to apoptotic, necrotic and mitotic cell death. The objectives of this study are to evaluate the use of ultrasound imaging and spectroscopy as a predictive marker of advanced tumour response to combined chemotherapy and radiotherapy. Since neoadjuvant treatments may also act on tumour vasculature to "normalize" it we will also evaluate blood-vessel imaging by standard Doppler-imaging and with standard higher-resolution imaging using clinically approved microbubble contrast agents.

The main goal, as described above, is to select the best ultrasound spectroscopy parameter to use as an early predictor of pathological complete response.

DETAILED DESCRIPTION:
We have previously demonstrated that high-frequency ultrasound and spectroscopy, and recently conventional-frequency ultrasound and spectroscopy may be used to detect cell death in vitro, in situ and in vivo. The method can detect different forms of cell death and has been demonstrated to be sensitive to apoptotic, necrotic and mitotic cell death. The objectives of this study are to evaluate the use of ultrasound imaging and spectroscopy as a predictive marker of advanced tumour response to combined chemotherapy and radiotherapy. Since neoadjuvant treatments may also act on tumour vasculature to "normalize" it we will also evaluate blood-vessel imaging by standard Doppler-imaging and with standard higher-resolution imaging using clinically approved microbubble contrast agents.

The main goal, as described above, is to select the best ultrasound spectroscopy parameter to use as an early predictor of pathological complete response.

Specifically, we will as a primary endpoint correlate changes in ultrasound backscatter parameters obtained throughout the course of treatment with pathological complete, partial, or complete and partial response. We ultimately hope to be able to generate a Receiver-Operator-Curve for each parameter beyond this pilot investigation. The ultrasound-spectroscopy parameters to be examined include mid-band fit, spectral-slope and histogram-distribution-fit parameters related to scatterer size and concentration. From these various receiver-operator curves the best ultrasound parameter for predicting response will be selected and will aid to define the clinical specificity and sensitivity of the technique.

The secondary endpoint in this study will include examining the change in size of the tumour, which will also be measured using conventional gold-standard B-scan ultrasound imaging (length by width by height in addition to volume) and correlating that to the spectroscopic ultrasound changes determined at different times during patient treatment.

Other secondary endpoints will include measuring changes in blood vessel distribution by standard Doppler-imaging and standard microbubble contrast agent imaging. As another secondary endpoint we will also correlate our ultrasound changes with 2 and 5-year long-term clinical outcome.

ELIGIBILITY:
INCLUSION CRITERIA:

The following criteria are necessary for study participation:

1. Histologically or cytologically confirmed breast carcinoma, stage I-IV, which has not been treated with any first-line therapy and will be treated with neoadjuvant chemotherapy or neoadjuvant combined chemo-radiotherapy.
2. Measurable disease by ultrasound, or MRI performed within 28 days prior to treatment.
3. Eastern Co-operative Oncology Group (ECOG) Performance Status of 0 or 1.
4. Life expectancy of at least 6 months.
5. Adequate bone marrow, liver and renal function as assessed by the following laboratory. Requirements to be conducted within 7 days prior to dosing:

   (i) hemoglobin >90 mg/dL (ii) leukocytes >3,000/mL (iii) absolute neutrophil count >1,500/mL (iv) platelets >100,000/mL (v) total bilirubin within normal institutional limits (vi) AST(SGOT)/ALT(SGPT) <2.5 X institutional upper limit of normal (vii) creatinine within normal institutional limits or creatinine clearance >60 mL/min/1.73 m2 for patients with creatinine levels above institutional upper limit of normal
6. Patients should have the ability to understand and the willingness to sign a written informed consent document. Signed informed consent must be obtained prior to any study specific procedures.

EXCLUSION CRITERIA

The following conditions will exclude women from participation:

1. Chemotherapy, radiotherapy, or major surgery within 4 weeks prior to registering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks prior to registration.
2. Receiving any other investigational agents.
3. Known brain metastases.
4. History of allergic reactions attributed to compounds of similar chemical or biologic composition.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Women who are receiving neoadjuvant chemotherapy or neoadjuvant chemo-radiotherapy for breast cancer.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2008-12-17 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
The primary Outcome will be correlate changes in ultrasound backscatter parameters obtained throughout the course of treatment with pathological complete, partial, or complete and partial response. | 2 and 5-year long-term clinical outcome
  Ultrasound spectroscopy parameters to be examined include mid-band fit parameters, spectral slope and histogram distribution fit parameters related to scatterer size and concentration. From these various receiver-operator curves, the best ultrasound parameter predictive response will be selected and will aid to define the clinical specificity and sensitivity of The technique.

SECONDARY OUTCOMES:
The secondary Outcome of this study will include examining the change in tumor size. | 2 and 5-year long-term clinical outcome
  The change in tumor size, which It will also be measured using conventional gold standard B-scan ultrasound images (length by width by height in addition to volume) and correlating it with spectroscopic ultrasound changes determined at different times during the patient's treatment.
Other secondary Outcome will include measuring changes in the blood vessels distribution in the tumor. | 2 and 5-year long-term clinical outcome
  Measurement of changes in the distribution of blood vessels according to the standard doppler-imaging and standard microbubbles contrast agent imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory J. Czarnota, Ph.D. M.D., Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada